CLINICAL TRIAL: NCT04537650
Title: The Pathophysiology of Swallowing Impairment in People Recovering From COVID-19
Brief Title: Swallowing Impairment After COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); McMaster University (Other); University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: CAPCR 20-5477; 3R01DC011020-08S1 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Swallowing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Ventilated: Participants who were diagnosed with COVID-19 prior to October, 2021 who required hospitalization in an ICU with mechanical ventilation during their illness.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VFSS)
- COVID-19 Non-Ventilated: Participants who were diagnosed with COVID-19 prior to October, 2021 who did not require mechanical ventilation during their illness.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Study (VFSS)

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic Swallowing Study (VFSS) — A standardized dynamic radiographic examination of oropharyngeal swallowing

SUMMARY:
This is an observational study, in which people recovering from COVID-19 infection will attend an outpatient clinic for a comprehensive swallowing assessment. The assessment will include a videofluoroscopy, measurement of respiratory-swallow coordination using a digital stethoscope, measures of tongue and cough strength and patient reported measures that will help us to understand the presence and impact of swallowing impairment (dysphagia) in this population.

DETAILED DESCRIPTION:
The recent spread of COVID-19 has led to an international pandemic, with >3 million confirmed cases to date worldwide, of which 1 million confirmed cases and >50,000 deaths have been reported in the USA. Infected individuals commonly experience severe respiratory difficulties and pneumonia, leading to hospital admission and the need for intensive care and mechanical ventilation. Emerging evidence suggests that impaired taste and smell may be early markers of the disease, and that in severe cases, there may be neurological damage in in the medulla, an important brainstem control site for both respiration and swallowing. Given the overlapping neuroanatomical regulation of breathing and swallowing, the investigators hypothesize that dysphagia (swallowing impairment) will be common in People recovering from COVID-19 (PrC-19) and associated with poorer outcomes.

The investigators will offer comprehensive swallowing assessments to PrC-19 after initial recovery and a confirmed negative test for continuing COVID-19 infection. Study sites will be located in the Toronto area (PI Steele); the Hamilton-Niagara region to the west of Toronto (Co-I Namasivayam-MacDonald) and in Gainesville, Florida (Co-I Plowman). The assessments will include the collection of case history information, videofluoroscopy (i.e., a dynamic swallowing x-ray), use of a digital stethoscope to measure respiratory-swallow coordination, measures of other risk factors for dysphagia (e.g. bulbar muscle strength) and patient-reported outcomes. Detailed analyses of the videofluoroscopy swallowing studies (i.e. dynamic x-rays) will identify specific measures of swallowing that fall outside the range of normal variation based on comparison to healthy reference values established through the PI's NIH-funded research program exploring swallowing physiology on liquids of different consistencies.

ELIGIBILITY:
Inclusion Criteria:

* People who tested positive or received a presumed positive diagnosis of COVID-19 infection not earlier than March 1, 2020 and who are at least 2 weeks post positive diagnosis and the initiation of medical management of COVID-19 infection
* Adequate comprehension of English to understand the consent form and follow study instructions

Exclusion Criteria:

* Age under 18 years old
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals recovering from COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- University of Florida, Gainesville, Florida, United States
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steele CM, Peladeau-Pigeon M, Barbon CAE, Guida BT, Namasivayam-MacDonald AM, Nascimento WV, Smaoui S, Tapson MS, Valenzano TJ, Waito AA, Wolkin TS. Reference Values for Healthy Swallowing Across the Range From Thin to Extremely Thick Liquids. J Speech Lang Hear Res. 2019 May 21;62(5):1338-1363. doi: 10.1044/2019_JSLHR-S-18-0448. PMID 31021676
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Steele CM, Bayley MT, Bohn MK, Higgins V, Peladeau-Pigeon M, Kulasingam V. Reference Values for Videofluoroscopic Measures of Swallowing: An Update. J Speech Lang Hear Res. 2023 Oct 4;66(10):3804-3824. doi: 10.1044/2023_JSLHR-23-00246. Epub 2023 Sep 5. PMID 37669617

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Ventilated: This group of participants were hospitalized and require ICU care with mechanical ventilation during their COVID-19 infection
- COVID-19 Non-ventilated: This group of participants did not require mechanical ventilation during their COVID-19 infection
Period: Overall Study
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Started | 8 | 36
Completed | 8 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- COVID-19 Ventilated: This was a group of Community-Dwelling adults who had a history of COVID-19 infection prior to October, 2021 and who were hospitalized and required ICU care with mechanical ventilation during their COVID-19 infection
- COVID-19 Non-ventilated: This was a group of Community-Dwelling adults who had a history of COVID-19 infection prior to October, 2021 but who did not require mechanical ventilation during their COVID-19 infection.
- Total: Total of all reporting groups
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated | Total
Number analyzed (Participants) | 8 | 36 | 44
Age, Continuous [Mean (Full Range); unit: years] | 62 [37 to 79] | 44 [21 to 78] | 48 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 30 | 31
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 34 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 33 | 38
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Taste or Smell Impairment [Count of Participants; unit: Participants] — Number of Participants reporting persisting taste or smell impairment at the time of data collection
  Participants
    YES (Taste/Smell impairment) | 7 | 13 | 20
    NO (No Taste/Smell impairment) | 1 | 23 | 24
SSQ [Median (Inter-Quartile Range); unit: units on a scale] — Score on the Sydney Swallow Questionnaire, a patient-reported dysphagia severity measure. Minimum possible score is 0. Maximum possible score is 1700. Scores > 234 are considered impaired. Higher scores indicate greater impairment. Population: Full Sydney Swallow Questionnare were missing for 12 participants in the non-ventilated and 2 participants in the ventilated group who reported no swallowing difficulties, and therefore did not complete the full questionnaire.
  units on a scale
    number analyzed (Participants) | 6 | 24 | 30
    (all) | 98 [52 to 303] | 232 [55 to 422] | 158 [56 to 396]
Time since diagnosis [Mean (Full Range); unit: Months] — Time (in months) since COVID-19 diagnosis at the point of data collection
  Months | 6 [2 to 14] | 7 [1 to 17] | 7 [1 to 17]
Tongue Weakness [Count of Participants; unit: Participants] — Number of participants displaying tongue weakness, defined as a 1-repetition-maximum anterior isometric pressure measure of < 40 kPa taken across 3 repeated maximum anterior isometric pressure measurements using the Iowa Oral Performance Instrument.
  Participants | 3 | 8 | 11
Reduced peak cough flow [Count of Participants; unit: Participants] — Reduced voluntary peak cough expiratory flow, defined as a peak cough flow measure < 270 l/s, measured using a mini-Wright analog peak-cough flow meter.
  Participants | 1 | 6 | 7
Fail water swallow screen (3 sips) [Count of Participants; unit: Participants] — Number of participants displaying overt signs of potential aspiration (coughs, throat clear, change of voice quality) on a water swallow screening test involving a series of 3 discrete comfortable sips of water.
  Participants | 4 | 14 | 18
Fail water swallow screen (90cc) [Count of Participants; unit: Participants] — umber of participants displaying overt signs of potential aspiration (coughs, throat clear, change of voice quality, or failure to complete task) on a water swallow screening test involving continuous drinking of 90cc of water.
  Participants | 3 | 13 | 16
SSQ Impaired [Count of Participants; unit: Participants] — Number of participants reporting self-perceived swallowing impairment at baseline defined as a score on the Sydney Swallow Questionnaire > 234. Population: Full Sydney Swallow Questionnare were missing for 12 participants in the non-ventilated and 2 participants in the ventilated group who reported no swallowing difficulties, and therefore did not complete the full questionnaire.
  Participants
    number analyzed (Participants) | 6 | 24 | 30
    (all) | 1 | 12 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Impaired Swallowing Safety
Description: Frequency of participants demonstrating airway invasion on thin liquids, defined as Penetration-Aspiration Scale score of 3 and higher (Rosenbek et al., 1996). Higher scores indicate worse function.
Time Frame: Videofluoroscopy session (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 3 | 1
Statistical Analysis 1: Comparison: COVID-19 Ventilated vs COVID-19 Non-ventilated; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 21, 95% CI 2-sided [1.8 to 243.24]

2. Primary Outcome: Number of Participants With Impaired Swallowing Efficiency
Description: Frequency of participants demonstrating pharyngeal residue on extremely thick liquids measured to fill more than 1.5% of an anatomical reference scalar [%(C2-4)squared] (Steele et al., 2019)
Time Frame: Videofluoroscopy session (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 4 | 0
Statistical Analysis 1: Comparison: COVID-19 Ventilated vs COVID-19 Non-ventilated; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 45, 95% CI 2-sided [4.15 to 487.5]

3. Secondary Outcome: Number of Participants With Prolonged Time-to-Laryngeal-Vestibule-Closure
Description: Frequency of participants displaying prolonged time to airway closure (i.e. Laryngeal Vestibule Closure) on thin liquids, defined as values falling above the healthy reference 75th percentile (Steele et al., 2023)
Time Frame: Videofluoroscopy session (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 6 | 14

4. Secondary Outcome: Number of Participants With Short Laryngeal Vestibule Closure Duration
Description: Frequency of participants displaying short airway closure (i.e. laryngeal vestibule closure) on thin liquids, defined as a duration below the healthy reference 25th percentile (Steele et al., 2023)
Time Frame: Videofluoroscopy session (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 3 | 4

5. Secondary Outcome: Number of Participants With Poor Pharyngeal Constriction
Description: Frequency of participants displaying poor pharyngeal constriction on extremely thick liquids, defined as pharyngeal area above the 75th percentile healthy reference value on the frame of maximum constriction (Steele et al., 2023)
Time Frame: Videofluoroscopy session (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 6 | 6

6. Secondary Outcome: Number of Participants With Impaired LVC Integrity
Description: Number of participants displaying incomplete laryngeal vestibule closure on thin liquids.
Time Frame: Videofluoroscopy (single timepoint only)
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
Number analyzed (Participants) | 8 | 36
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Within 1 week of data collection
Arm/Group | COVID-19 Ventilated | COVID-19 Non-ventilated
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/36
Other Adverse Events (participants affected / at risk) | 0/8 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04537650/Prot_SAP_000.pdf